CLINICAL TRIAL: NCT05702229
Title: An Open-Label, Multi-Drug, Multi-Centre, Phase II Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Novel Combinations in Participants With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Novel Combinations in Participants With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7986C00001; 2022-002840-29 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2023-01-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: Locally advanced; Metatstatic; Gastric adenocarcinoma; GEJ adenocarcinoma; GEMINI-Gastric
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol; XELOX; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Substudy 1 (Experimental): Volrustomig plus XELOX (oxaliplatin and capecitabine) or FOLFOX (oxaliplatin and 5-FU/CF)
  Interventions: Drug: Volrustomig; Drug: FOLFOX; Drug: XELOX
- Substudy 2 (Experimental): Rilvegostomig plus XELOX (oxaliplatin and capecitabine) or FOLFOX (oxaliplatin and 5-FU/CF)
  Interventions: Drug: Rilvegostomig; Drug: FOLFOX; Drug: XELOX
- Substudy 3 (Experimental): AZD0901 plus volrustomig and 5-fluorouracil or capecitabine
  Interventions: Drug: Volrustomig; Drug: AZD0901; Drug: 5-Fluorouracil; Drug: Capecitabine
- Substudy 4 (Experimental): AZD0901 plus rilvegostomig and 5-fluorouracil or capecitabine
  Interventions: Drug: Rilvegostomig; Drug: AZD0901; Drug: 5-Fluorouracil; Drug: Capecitabine
- Substudy 5 (Experimental): AZD7789 plus XELOX (oxaliplatin and capecitabine) or FOLFOX (oxaliplatin and 5-FU/CF)
  Interventions: Drug: FOLFOX; Drug: XELOX; Drug: AZD7789
- Substudy 6 (Experimental): AZD0901 plus AZD7789 and 5-fluorouracil or capecitabine
  Interventions: Drug: AZD7789; Drug: AZD0901; Drug: 5-Fluorouracil; Drug: Capecitabine

INTERVENTIONS:
Drug: Rilvegostomig — an anti PD-1 and anti-TIGIT bispecific antibody; IV infusion
  Arms: Substudy 2; Substudy 4
Drug: Volrustomig — an anti PD-1 and anti CTLA-4 bispecific antibody; IV infusion
  Arms: Substudy 1; Substudy 3
Drug: FOLFOX — 5-fluorouracil 400 mg/m^2 IV, oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2 (or levoleucovorin 200 mg/m^2 when locally preferred and available), day 1, 5-fluorouracil 1200 mg/m^2 IV 24 h day 1-2
  Arms: Substudy 1; Substudy 2; Substudy 5
Drug: XELOX — capecitabine 1000 mg/m^2 BID, days 1 to 14, oxaliplatin 130 mg/m^2, day 1
  Arms: Substudy 1; Substudy 2; Substudy 5
Drug: AZD7789 — an anti PD 1 and anti TIM 3 bispecific antibody; IV infusion
  Arms: Substudy 5; Substudy 6
Drug: AZD0901 — an anti Claudin18.2 ADC; IV infusion
  Arms: Substudy 3; Substudy 4; Substudy 6
Drug: 5-Fluorouracil — 5-FU, IV infusion, Q3W
  Arms: Substudy 3; Substudy 4; Substudy 6
Drug: Capecitabine — Oral take, Q3W
  Arms: Substudy 3; Substudy 4; Substudy 6

SUMMARY:
This is a Phase II, open-label, multi-drug, multi-centre study designed to assess the efficacy, safety, tolerability, pharmacokinetics, and immunogenicity of novel combination therapies in participants with locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma.

DETAILED DESCRIPTION:
Approximately 240 participants will be assigned across 6 substudies, with approximately 40 evaluable participants of the confirmed recommend dose by SRC for study intervention in each corresponding substudy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of signing the ICF.
* Body weight > 35 kg.
* Previously untreated for unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.
* Has measurable target disease assessed by the Investigator based on RECIST 1.1.
* ECOG PS zero or one.
* Life expectancy of at least 12 weeks.
* Adequate organ and bone marrow function.
* Has central lab confirmed Claudin18.2 status at screening from archival tumour collected within past 24 months or from a fresh biopsy when Substudy 3, Substudy 4 or Substudy 6 is open for recruitment.

Exclusion Criteria:

* Participants with HER2-positive (3+ by IHC, or 2+ by IHC and positive by in situhybridisation) or indeterminate gastric or GEJ carcinoma.
* Untreated or progressive CNS metastatic disease, any leptomeningeal disease, or cord compression.
* Participants with ascites which cannot be controlled with appropriate interventions.
* Active infectious diseases, including tuberculosis, HIV infection, or hepatitis A/B/C.
* Uncontrolled intercurrent illness.
* Active or prior documented autoimmune or inflammatory disorders requiring systemic treatment with steroids or other immunosuppressive treatment.
* History of another primary malignancy.
* Previous treatment with an immune-oncology agent.
* Previous treatment with any modalities of Claudin18.2 target therapy or MMAE exposure (when Substudy 3, Substudy 4, or Substudy 6 is open for recruitment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
ORR (per RECIST 1.1 as assessed by Investigator) | Through substudy completion, an average of 2 years
  the proportion of participants who have a confirmed complete response or confirmed partial response, as determined by the Investigator at local site per RECIST 1.1.
PFS6 (per RECIST 1.1 as assessed by Investigator) | Through substudy completion, an average of 2 years
  the proportion of participants alive and progression-free at 6 months.

SECONDARY OUTCOMES:
PFS per RECIST 1.1 as assessed by the Investigator | Through substudy completion, an average of 2 years
  the time from the start of study intervention until progression per RECIST 1.1 as assessed by the Investigator at the local site or death due to any cause in the absence of progression.
OS | Through substudy completion, an average of 2 years
  the time from the start of study intervention until the date of death due to any cause.
other safety related endpoints | Through substudy completion, an average of 2 years
  Incidence of AEs, AESIs, and SAEs.
DoR per RECIST 1.1 based on Investigator assessment. | Through substudy completion, an average of 2 years
  the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 by the Investigator at local site or death due to any cause in the absence of disease progression.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Grand Rapids, Michigan
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, The Bronx, New York
  - Research Site, Pittsburgh, Pennsylvania
- China (8):
  - Research Site, Beijing
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Wuhan
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Sunto-gun
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Elche(Alicante)
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Santander
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Edinburgh
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home